CLINICAL TRIAL: NCT04804930
Title: Prognostic Value of Trichoscopy in Patients With Systemic Scleroderma
Brief Title: Trichoscopy and Systemic Scleroderma
Acronym: TRICHLOSCLERO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_87; 2020-A00566-33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Scleroderma, Systemic
Keywords: Trichoscopy; Dermoscopy; Systemic Scleroderma; Scalp
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with systemic scleroderma
  Interventions: Procedure: picture
- healthy subject: healthy subject without systemic scleroderma or known hair or scalp disease
  Interventions: Procedure: picture

INTERVENTIONS:
Procedure: picture — We will perform a non-invasive assessment of the scalp with a dermoscope by taking two standardized pictures on the frontal area and the occipital area in order to a blinded analysis of trichoscopic patterns
  Other Names: Non-invasive trichoscopy: dermoscopic assessment of the scalp (picture)

SUMMARY:
* Few data are available on scalp involvement in systemic scleroderma.
* Few data are available on the association between scalp abnormalities and features of systemic scleroderma
* Trichoscopy is a simple, reproducible, noninvasive examination that is part of the examination of hairy areas in routine dermatologic practice
* There is a lack of simple, noninvasive examinations to evaluate patients with systemic scleroderma

The objective will be to evaluate the contribution of trichoscopy in the evaluation of patients with systemic scleroderma

ELIGIBILITY:
Inclusion Criteria:

* Patient who fulfils the Systemic scleroderma ACR-EULAR 2013 criteria
* Signed informed consent
* Being social insured

Exclusion Criteria:

* Patients aged less than 18 years old
* patients under legal protection
* patients deprived of their liberty
* patients in emergency situations
* patients who refused or unable to give informed consent
* For the control group: sclap inflammatory disease active the day of the examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with systemic scleroderma
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of elementary lesions observed by trichoscopic assessment of the scalp | Baseline
  Comparison of the frequencies of elementary lesions visualized in patients with systemic scleroderma and healthy subjects

SECONDARY OUTCOMES:
Correlation between visceral damage of systemic scleroderma and trichoscopic features | Baseline
  Frequency of visceral damage of systemic scleroderma: pulmonary hypertension, lung fibrosis, kidney failure.
Correlation between global severity of systemic scleroderma and trichoscopic features | Baseline
  Correlation between EUSTAR score, Rodnan score, Medsger's score and trichoscopic features
Correlation between autoimmune profile of sclerodermic patients and trichoscopic features | Baseline
  Correlation of antibodies, inflammatory profile of patients with trichoscopic features.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Sobanski, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France